CLINICAL TRIAL: NCT03804684
Title: How Does the visuALL Field Analyzer (vFA) Compare to Standard Automatic Perimetry (SAP) in Patients With Mild and Moderate Chronic Open Angle Glaucoma (COAG) and Subjects Without Eye Problems?
Brief Title: visuALL Field Analyzer (vFA) Compared to Standard Humphrey Automated Perimetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Olleyes, Inc. (Industry)
Responsible Party: Principal Investigator, M. Reza Razeghinejad MD, Principal Investigator, Wills Eye
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB Control #18-768E
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Glaucoma, Open-Angle
Keywords: open angle glaucoma; visual field; Standard Automatic Perimetry
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy Controls (Experimental): Healthy subjects between 21 and 80 years of age with no eye diseases (normal appearing optic nerve and retina, intraocular eye pressure less than 19 millimeters of mercury, normal and reliable standard automatic perimetry, and spherical refraction less than 3 diopters and cylinder correction equal to 2 diopters or less. All subjects will perform Standard Automatic Perimetry Humphrey Field Analyzer and visuALL Field Analyzer to measure peripheral and central visual field.
  Interventions: Diagnostic Test: Standard Automatic Perimetry Humphrey Field Analyzer; Diagnostic Test: visuALL Field Analyzer
- Mild and Moderate Glaucoma (Experimental): Subjects between 21 and 80 years of age with Mild or Moderate Glaucoma. Eyes will have a reliable standard automatic perimetry with no more than -6 mean deviation (Mild) and between -6 mean and -12 mean deviation (Moderate). Spherical refraction will be less than 3 diopters and cylinder correction equal to 2 diopters or less. All subjects will perform Standard Automatic Perimetry Humphrey Field Analyzer and visuALL Field Analyzer to measure peripheral and central visual field.
  Interventions: Diagnostic Test: Standard Automatic Perimetry Humphrey Field Analyzer; Diagnostic Test: visuALL Field Analyzer

INTERVENTIONS:
Diagnostic Test: Standard Automatic Perimetry Humphrey Field Analyzer — Standard Automatic Perimetry (SAP) Humphrey Field Analyzer (HFA) 24-2, Swedish Interactive Threshold Algorithm (SITA) Standard Strategy measures peripheral and central vision in an ophthalmic setting.
  Other Names: SAP HFA
Diagnostic Test: visuALL Field Analyzer — visuALL Field Analyzer a new portable hardware and software virtual reality system measures peripheral and central vision to improve early detection of glaucoma damage in a non ophthalmic setting.
  Other Names: vFA

SUMMARY:
To determine age-adjusted reference values of the visuALL Field Analyzer (vFA) retinal sensitivity and to assess the repeatability of the measured values and compare them with those measured by a Standard Automatic Perimetry (SAP).

DETAILED DESCRIPTION:
Standard Automatic Perimetry (SAP) is the gold standard test for the evaluation of central and peripheral retinal sensitivity to light for detection and monitoring optic nerve diseases such as glaucoma. The current device has its own limitation such as positioning for the duration of the test which makes is hard for older patients especially those with back or other musculoskeletal diseases, artifact of the corrective lenses used to accommodate the patients refractive errors, etc.

Several devices have been developed since the advent of the Octopus Perimeter 3-5 and the Humphrey Field Analyzer (HFA), in an effort to improve the test reliability and patient comfort.

The main goal of this study is to evaluate the repeatability of a novel psychophysical platform that takes advantage of a Head Mounted Device (HMD) with eye tracking capabilities. Other objectives of this study include the development of an initial reference database and comparison of the measured parameters with HFA.

ELIGIBILITY:
Inclusion Criteria:

* age 21 to 80 years
* Healthy subjects with no eye diseases, normal appearing optic nerve and retina, intraocular pressure less than 19 millimeters mercury and normal standard automatic perimetry (SAP).
* mild glaucoma subjects with less than -6 mean deviation
* moderate glaucoma subjects with -6 to -12 mean deviation

Exclusion Criteria:

* spherical refraction outside ± 3.0 diopters and cylinder correction outside 2.0 diopters
* Unreliable SAP (false positives, fixation losses and false negatives greater than 25% and/or observable testing artifacts)
* Unreliable visuALL Field Analyzer (vFA) (greater than 25% false positive, excessive fixation losses)
* SAP abnormality with pattern loss consistent with neurologic and/or other ocular diseases than glaucoma
* Intraocular surgery in study eye (except non-complicated cataract or refractive surgery performed more than 6 months before enrollment and without posterior capsule opacification)
* History of systemic condition known to affect visual function
* History of medication known to affect visual function

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Reza Razeghinejad, MD, Principal Investigator — Wills Eye
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Razeghinejad R, Gonzalez-Garcia A, Myers JS, Katz LJ. Preliminary Report on a Novel Virtual Reality Perimeter Compared With Standard Automated Perimetry. J Glaucoma. 2021 Jan 1;30(1):17-23. doi: 10.1097/IJG.0000000000001670. PMID 32941320

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Glaucoma patients with mild or moderate visual field loss and subjects with healthy vision were enrolled to form two groups for comparison of two methods of visual field testing. Subjects unable to perform testing or test reliability did not meet inclusion criteria in 3 of the Healthy Controls and 18 of the Glaucoma Group. Therefore, 21 participants were excluded from results.
Groups:
- Healthy Controls: Healthy subjects between 21 and 80 years of age with no eye diseases. Eyes will have normal appearing optic nerve and retina, intraocular eye pressure less than 19 millimeters of mercury, normal, reliable standard automatic perimetry and spherical refraction less than 3 diopters and cylinder correction equal to 2 diopters or less. All subjects will perform Standard Automatic Perimetry Humphrey Field Analyzer and visuALL Field Analyzer to measure peripheral and central visual field.
- Glaucoma Group: Subjects between 21 and 80 years of age with Mild or Moderate Glaucoma. Eyes will have reliable standard automatic perimetry with no more than -6 mean deviation (mild glaucoma) and between -6 mean and -12 mean deviation (moderate glaucoma); and spherical refraction less than 3 diopters and cylinder correction equal to 2 diopters or less. All subjects will perform Standard Automatic Perimetry Humphrey Field Analyzer and visuALL Field Analyzer to measure peripheral and central visual field.
Period: Overall Study
Arm/Group | Healthy Controls | Glaucoma Group
Started | 28 | 44
Completed | 25 | 26
Not Completed | 3 | 18
Not completed — Subjects unable to perform testing or test reliability did not meet inclusion criteria. | 3 | 18

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Glaucoma Group: Subjects between 21 and 80 years of age with Mild and Moderate Glaucoma. Eyes will have reliable standard automatic perimetry with no more than -6 mean deviation (mild glaucoma) and between -6 mean and -12 mean deviation (moderate glaucoma); and spherical refraction less than 3 diopters and cylinder correction equal to 2 diopters or less. All subjects will perform Standard Automatic Perimetry Humphrey Field Analyzer and visuALL Field Analyzer to measure peripheral and central visual field.
  Standard Automatic Perimetry Humphrey Field Analyzer: Standard Automatic Perimetry (SAP) Humphrey Field Analyzer (HFA) 24-2, Swedish Interactive Threshold Algorithm (SITA) Standard Strategy measures peripheral and central vision in an ophthalmic setting.
  visuALL Field Analyzer: visuALL Field Analyzer a new portable hardware and software virtual reality system measures peripheral and central vision to improve early detection of glaucoma damage in a non ophthalmic setting.
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Glaucoma Group | Total
Number analyzed (Participants) | 28 | 44 | 72
Number analyzed (Eyes) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 23 | 43
  >=65 years | 8 | 21 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 10 | 23 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 25 | 44 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 24 | 34
  White | 17 | 20 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 44 | 72
Mild to Moderate Glaucoma [Count of Participants; unit: Participants] | 0 | 44 | 44
Number of eyes analyzed [Number; unit: number of eyes]
  total eyes analyzed | 50 | 52 | 102
  eyes with mild visual field defects | 0 | 36 | 36
  eyes with moderate visual field defects | 0 | 13 | 13
  eyes with severe visual field defects | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Retinal Sensitivity From Two Machines
Description: Mean (Average) retinal sensitivity to light as measured in decibels in multiple spots across the central and peripheral retina (entire visual field). Higher numbers translate to dimmer light which when detected means better vision.
Time Frame: three hours
Measure: Mean (Standard Deviation); unit: decibels
Units Other Than Participants: Eyes
Groups:
- Healthy Controls: Healthy subjects between 21 and 80 years of age with no eye diseases. Fifty eyes with normal appearing optic nerve and retina, intraocular eye pressure less than 19 millimeters of mercury, normal, reliable standard automatic perimetry and spherical refraction less than 3 diopters and cylinder correction equal to 2 diopters or less. All subjects performed Standard Automatic Perimetry Humphrey Field Analyzer and visuALL Field Analyzer to measure peripheral and central visual field.
- Glaucoma Group: Subjects between 21 and 80 years of age with Mild and Moderate Glaucoma. Fifty-two eyes with reliable standard automatic perimetry with no more than -6 mean deviation (mild glaucoma) and between -6 mean and -12 mean deviation (moderate glaucoma); and spherical refraction less than 3 diopters and cylinder correction equal to 2 diopters or less. All subjects performed Standard Automatic Perimetry Humphrey Field Analyzer and visuALL Field Analyzer to measure peripheral and central visual field.
Arm/Group | Healthy Controls | Glaucoma Group
Number analyzed (Participants) | 25 | 26
Number analyzed (Eyes) | 50 | 52
decibels
  Global field from Humphrey Visual Field | 29.9 (1.4) | 24.8 (3.9)
  Global field from VisuALL | 28.7 (1.3) | 22.9 (4.9)
  Inferior nasal quadrant from Humphrey Visual Field | 30.3 (1.3) | 24.8 (5.8)
  Inferior nasal quadrant from VisuALL | 28.7 (1.6) | 23.3 (6.9)
  Superior hemifield from Humphrey Visual Field | 29.5 (1.5) | 23.7 (5.0)
  Superior hemifield from VisuALL | 28.6 (1.6) | 21.8 (6.5)

2. Primary Outcome: Global Correlation (Agreement Between Two Machines in the Overall Visual Field)
Description: Correlation (Agreement) between Humphrey Visual Field and VisuALL retinal sensitivity as measured by mean deviation (light measurement in decibels) in multiple spots across the central and peripheral retina (entire visual field). This is the amount of agreement of the measure threshold, which is the lowest level of light detected in different points across the visual field (overall), between two testing machines.
Time Frame: three hours
Population: The overall mean retinal sensitivity (lowest level of light detected) measured by two perimetry machines was compared in both normal and glaucoma subjects. This is the difference between the results of the two machines for healthy and glaucoma eyes across their visual field (overall).
Measure: Mean (1% Confidence Interval); unit: decibels
Units Other Than Participants: Eyes
Groups:
- Glaucoma Group: Subjects between 21 and 80 years of age with Mild and Moderate Glaucoma. Eyes will have reliable standard automatic perimetry with no more than -6 mean deviation (mild glaucoma) and between -6 mean and -12 mean deviation (moderate glaucoma); and spherical refraction less than 3 diopters and cylinder correction equal to 2 diopters or less. All subjects will perform Standard Automatic Perimetry Humphrey Field Analyzer and visuALL Field Analyzer to measure peripheral and central visual field.
Arm/Group | Healthy Controls | Glaucoma Group
Number analyzed (Participants) | 25 | 26
Number analyzed (Eyes) | 50 | 52
decibels | 0.5 [0 to 1] | 0.8 [0 to 1]

3. Secondary Outcome: Inferior Nasal Quadrant Correlation (Agreement Between Two Machines in the Inferior Nasal Visual Field)
Description: Correlation (Agreement) between Humphrey Visual Field and VisuALL retinal sensitivity as measured by mean deviation (light measurement in decibels) in multiple spots across the inferior nasal visual field. This is the amount of agreement of the measure threshold, which is the lowest level of light detected in different points across the inferior (lower) nasal portion of the visual field, between two testing machines.
Time Frame: three hours
Population: The overall mean retinal sensitivity (lowest level of light detected) measured by two perimetry machines was compared in both normal and glaucoma subjects. This is the difference between the results of the two machines for healthy and glaucoma eyes across their inferior nasal visual field).
Measure: Mean (1% Confidence Interval); unit: decibels
Units Other Than Participants: Eyes
Arm/Group | Healthy Controls | Glaucoma Group
Number analyzed (Participants) | 25 | 26
Number analyzed (Eyes) | 50 | 52
decibels | 0.3 [0 to 1] | 0.8 [0 to 1]

4. Secondary Outcome: Superior Hemifield Correlation (Agreement Between Two Machines in the Superior Hemifield Visual Field
Description: Correlation (Agreement) between Humphrey Visual Field and VisuALL retinal sensitivity as measured by mean deviation (light measurement in decibels) in multiple spots across the superior (upper) hemifield portion of the visual field. This is the amount of agreement of the measure threshold, which is the lowest level of light detected in different points across the visual field in the superior hemifield, between two testing machines.
Time Frame: three hours
Population: The mean retinal sensitivity (lowest level of light detected) measured by two perimetry machines was compared in both normal and glaucoma subjects. This is the difference between the results of the two machines for healthy and glaucoma eyes across the superior hemifield portion of their visual field.
Measure: Mean (1% Confidence Interval); unit: decibels
Units Other Than Participants: Eyes
Arm/Group | Healthy Controls | Glaucoma Group
Number analyzed (Participants) | 25 | 26
Number analyzed (Eyes) | 50 | 52
decibels | 0.4 [0 to 1] | 0.6 [0 to 1]

ADVERSE EVENTS:
Time Frame: 3 hours
Arm/Group | Healthy Controls | Glaucoma Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/44
Other Adverse Events (participants affected / at risk) | 0/28 | 0/44

LIMITATIONS AND CAVEATS:
Disadvantages of VisuALL are similar to standard automated perimetry. They rely on patient cooperation and concentration during visual field examination. In addition, the system does not include follow-up analysis. The head-mounted device may not be preferred by subjects with claustrophobic tendencies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03804684/Prot_SAP_000.pdf